CLINICAL TRIAL: NCT04990219
Title: Interventional, Randomized, Double-blind, Placebo-controlled, Parallel-group, Phase 1B Study Investigating the Effects of Lu AG06466 for the Treatment of Spasticity in Patients With Multiple Sclerosis
Brief Title: A Study of Lu AG06466 for the Treatment of Spasticity in Participants With Multiple Sclerosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated for strategic reasons
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19366A; 2021-001230-18 (EudraCT Number)
Record Dates: First submitted 2021-07-29; First posted 2021-08-04 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lu AG06466 (Experimental): Participants will receive Lu AG06466 at a starting dose orally once daily for 4 days (Day 1 to Day 4), followed by Lu AG06466 at a higher titrated dose orally once daily for 4 days (Day 5 to Day 8), followed by Lu AG06466 at a higher titrated treatment dose orally once daily from Day 9 until Day 35/Week 5.
  Interventions: Drug: Lu AG06466
- Placebo (Placebo Comparator): Participants will receive Lu AG06466-matching placebo orally once daily until Day 35/Week 5.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lu AG06466 — Lu AG06466 - capsule
  Arms: Lu AG06466
Drug: Placebo — Placebo - capsule
  Arms: Placebo

SUMMARY:
The main purpose of this study is to investigate Lu AG06466 as a treatment for spasticity in participants with multiple sclerosis (MS).

DETAILED DESCRIPTION:
The participants will be randomized to Lu AG06466 or placebo in a 2:1 ratio.

ELIGIBILITY:
Key Inclusion Criteria:

* The participant has a diagnosis of MS, as per the 2017 McDonald criteria.
* The participant has clinically stable MS (such as no relapse and/or stable Expanded Disability Status Scale [EDSS] or alternative clinical assessment score) for at least 6 months prior to screening.
* The participant has ongoing spasticity for at least 90 days prior to screening.
* The participant is on a stable regimen for at least 30 days prior to screening for all medications and non pharmacological therapies, including therapies that are intended to alleviate spasticity (for example, oral baclofen, tizanidine, dalfampridine), and willing to remain on the same regimen throughout the duration of the study.
* The participant reports walking impairment due to lower limb spasticity.

Key Exclusion Criteria:

* The participant has any concomitant disease or disorder that has spasticity-like symptoms or that may influence the participant's level of spasticity or the participant's overall ability to participate in the study.
* The participant has ambulation difficulties due to any concomitant disease or disorder other than MS.
* The participant has any known or suspected hypersensitivity to cannabinoids (CBs) or any of the excipients of the investigational medicinal product (IMP).
* The participant has a positive drug screening test, except for non-CB medications used to treat a medical condition and reported as such by the participant; the participant has a positive drug screen test for cannabis/delta-9-tetrahydrocannabinol.

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Spasticity Response | Baseline to Week 5
  Spasticity response defined as ≥30% increase from baseline in spasticity Numerical Rating Scale (NRS) score
Change from Baseline to Week 5 in Spasticity NRS Score | Baseline, Week 5

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (7):
- United States (4):
  - Mountain View Clinical Research, Denver, Colorado
  - Johns Hopkins University, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Wake Research - Clinical Research Center of Nevada, Las Vegas, Nevada
- Germany (3):
  - Universitätsklinikum Düsseldorf, Dusseldorf NRW
  - Neurostimulation Center for Movement Disorders, Mainz
  - Center of Neurology, Hertie Institute for Clinical Brain Research, Tübingen